CLINICAL TRIAL: NCT06224582
Title: Efficacy and Safety of Yinxingmihuan Oral Solution in Treatment of Chest Pain After PCI: A Multicenter, Prospective, Randomized, Double-blind, Placebo-Controlled Study
Brief Title: Yinxingmihuan Oral Solution in Treatment of Chest Pain After PCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Yinxingmihuan01
Record Dates: First submitted 2024-01-16; First posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2021-03

CONDITIONS: Chronic Stable Angina
MeSH Terms: conditions — Angina, Stable | interventions — Ginkgo biloba extract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yinxingmihuan group (Experimental): standardized medical treatment regimen plus Yinxingmihuan oral solution (oral, 10 ml once, 3 times a day)
  Interventions: Drug: Yinxingmihuan oral solution
- Placebo group (Placebo Comparator): standardized medical treatment regimen plus Placebo oral solution (oral, 10 ml once, 3 times a day)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Yinxingmihuan oral solution — Yinxingmihuan oral solution is made of Ginkgo leaf extract and armillariella mellea powders.
  Other Names: Ginkgo leaf extract and armillariella mellea powders
  Arms: Yinxingmihuan group
Drug: Placebo — The placebo oral solution is in the same appearance, color, smell and taste as the experimental Yinxingmihuan oral solution.
  Arms: Placebo group

SUMMARY:
A prospective, multi-center, double-blind, randomized, placebo-controlled trial is conducted to evaluate the efficacy and safety of Yinxingmihuan oral solution in the treatment of chest pain after percutaneous coronary intervention (PCI) in patients with stable angina. Patients should undergo at least 1-week standardized medical treatment phase before randomization. The primary end point is the 12-week angina frequency assessed on the basis of Seattle Angina Questionnaire (SAQ) subscales. The main secondary endpoint is the improvement of anxiety assessed by Hamilton Anxiety Scale (HAMA) to evaluate its effectiveness for chest pain caused by psychological factors.

ELIGIBILITY:
Inclusion Criteria:

* male or female aged 18-85 years;
* patients with a history of percutaneous coronary intervention for coronary heart disease for more than 30 days and less than 180 days, without need of further elective coronary revascularization (PCI, CABG) judged by cardiovascular specialists;
* patients with symptoms such as chest distress, chest pain, palpitation, pain in shoulder and back, shortness of breath, weakness, activity intolerance, etc. Angina frequency (AF) score in Seattle Angina Questionnaire (SAQ) no more than 80;
* Hamilton Anxiety Scale score between 7 and 21 (mild to moderate anxiety);
* written informed consent.

Exclusion Criteria:

* women who are pregnant or preparing to be pregnant or nursing, menstruating women;
* women of child-bearing age who do not agree to use contraception during the medication phase;
* patients with severe anxiety (Hamilton Anxiety Scale score more than 21);
* patients with severe depression (Hamilton Depression Scale score not less than 24);
* patients who are currently taking anti-anxiety drug;
* participants with stable angina classified into Canadian Cardiovascular Society (CCS) Grade 4;
* uncontrolled hypertension (systolic > 180 mmHg or diastolic > 100 mmHg) despite using ongoing antihypertensive treatment;
* heart failure assessed by New York Heart Association (NYHA);
* patients with coronary heart disease and atrial fibrillation;
* clinically significant complications, including liver dysfunction (ALT or AST level more than 2 times higher than normal), renal dysfunction (serum creatinine level more than 2 times higher than normal), severe cardiopulmonary dysfunction, pulmonary hypertension, chronic obstructive pulmonary disease, history of cerebral hemorrhage or epilepsy, with need of anticonvulsant drugs;
* within 7 days of introduction period, patients who no longer have angina-related symptoms;
* within the three months before start of the study, patients with myocardial infarction or CCS 4 angina;
* patients with acute coronary syndrome confirmed by examinations and other chest pain caused by rheumatic heart disease, dilated cardiomyopathy, severe neurosis, menopausal syndrome, hyperthyroidism, cervical spondylosis, bilio-cardiac syndrome, gastroesophageal reflux, hiatal hernia, aortic dissection, pulmonary embolism, mediastinal hematoma, etc;
* history of specific bleeding or bleeding caused by warfarin;
* patients with previous hematopoietic diseases;
* patients who have undergone surgery (not including PCI) within the last 4 weeks and are prone to bleeding;
* patients who participate in any other clinical study or take any other investigational drug within 90 days;
* patients who are known or suspected to be allergic to the drug in this study or are allergic constitution;
* drug abusers who have a history of alcohol abuse or drug dependence in the past 2 years;
* psychopath;
* patients who have been judged by their doctors to be ineligible for the study;
* patient who is a family member or relative of the staff working in the centers.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2020-12-30 (Actual); Primary Completion 2023-12-25 (Actual); Study Completion 2023-12-25 (Actual)

PRIMARY OUTCOMES:
SAQ-angina frequency | at 12-week follow-up
  angina frequency assessed on the basis of Seattle Angina Questionnaire (SAQ-AF)

SECONDARY OUTCOMES:
HAMA improvement | at 12-week follow-up
  variation of the value of Hamilton Anxiety Scale (HAMA) at 12-week follow-up compared with baseline
CCS grade | before randomization, in 4,8,12,16 and 20 weeks
  angina grade assessed by Canadian Cardiovascular Society (CCS)
NYHA class | before randomization, in 4,8,12,16 and 20 weeks
  heart function assessed by New York Heart Association (NYHA)
VAS | before randomization, in 4,8,12,16 and 20 weeks
  generic health status assessed by visual analogue scale (VAS)
HAMA reductive ratio | at 12-week follow-up
  variation of Hamilton Anxiety Scale (HAMA) score at 12-week follow-up compared with baseline divided by the baseline value
HAMD depression score | before randomization, in 4,8,12,16 and 20 weeks
  proportion of participants with improvement or disappear of depression according to Hamilton Depression Scale (HAMD)
weekly angina frequency | before randomization, in 4,8,12,16 and 20 weeks
  weekly angina frequency recorded by the participants' diary cards
SF-12 score | before randomization, in 4,8,12,16 and 20 weeks
  generic health status measured by 12-Item Short Form Health Survey (SF-12)
Nitroglycerin discontinuation rate | before randomization, in 4,8,12,16 and 20 weeks
  proportion of participants that no longer need any nitroglycerin medications

OTHER OUTCOMES:
SAQ-PL | before randomization, in 4,8,12,16 and 20 weeks
  Physical limitation assessed on the basis of Seattle Angina Questionnaire
SAQ-AS | before randomization, in 4,8,12,16 and 20 weeks
  Anginal stability assessed on the basis of Seattle Angina Questionnaire
SAQ-TS | before randomization, in 4,8,12,16 and 20 weeks
  Treatment satisfaction assessed on the basis of Seattle Angina Questionnaire
SAQ-DP | before randomization, in 4,8,12,16 and 20 weeks
  Disease perception assessed on the basis of Seattle Angina Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital, National Center for Cardiovascular Diseases，Chinese Academy of Medical Sciences, Beijing, China